CLINICAL TRIAL: NCT04537507
Title: Is Atrial Fibrillation is Associated With Non-significant Coronary Angiography Findings?
Brief Title: Atrial Fibrillation and Non-obstructive Coronary Lesions
Acronym: AF-CAD
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other); Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Lukasz Kuzma, Principal Investigator, Medical University of Bialystok
Other Study IDs: UMB-KKI-102
Record Dates: First submitted 2020-08-22; First posted 2020-09-03 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-09

CONDITIONS: Fibrillation, Atrial; Coronary Artery Disease; Chronic Kidney Diseases
Keywords: Fibrillation, Atrial; Coronary Artery Disease; Chronic Kidney Disease
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent coronary angiography: We reviewed medical notes of patients hospitalized for coronary angiography because of exacerbated angina (recurrent chest pain, classical stable angina, long history of chest pain/angina or other symptoms such as dyspnea). We excluded patients with acute coronary syndromes (ACS), Tako-tsubo cardiomiopathy and history of ischemic heart disease, as well as those referred for coronary angiography before heart valve surgery. Prior cardiosurgical valve replacement was also the exclusion criterion.
  Interventions: Procedure: Coronary angiography

INTERVENTIONS:
Procedure: Coronary angiography

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia associated with excessive risk of ischemic stroke and heart failure as well as reduced life expectancy. On the other hand, chronic coronary syndromes (CCS) remains the main cause of morbidity and mortality in an aging population. Both disease entities share common risk factors such as hypertension, diabetes and obesity The purpose of the study is to investigate the hypothesis indicating lack of significant coronary lesions in AF vs. sinus rhythm (SR) patients.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) and chronic coronary syndromes (CCS) share common risk factors and both disease entities frequently co-exist. Additionally, AF symptoms may mimic CCS. Objectives: To investigate the hypothesis indicating lack of significant coronary lesions in AF vs. sinus rhythm (SR) patients.

The prevalence of CCS in patients with AF varies from 17% to 47% whereas AF in patients with CCS is much less common, ranging from 0.2% to 5.Patients with AF more often have concomitant CCS as compared with sinus rhythm controls. Additionally, AF is more frequently present in patients with either peripheral- or cerebrovascular artery disease than in non-atherosclerotic individuals We conducted a multi-center retrospective study including consecutive patients referred for elective coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Coronary angiography

Exclusion Criteria:

* We excluded patients with acute coronary syndromes (ACS), Tako-tsubo cardiomiopathy and history of ischemic heart disease, as well as those referred for coronary angiography before heart valve surgery. Prior cardiosurgical valve replacement was also the exclusion criterion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We conducted a multi-center retrospective study including consecutive patients referred for elective coronary angiography.
Sampling Method: Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Coronary artery disease | Through study completion, an average of 8 years
  Number of Participants with significant findings on coronary angiography

CONTACTS AND LOCATIONS:
Locations (5):
- Poland (3):
  - Department of Cardiology, Medical University of Bialystok, Bialystok, Poland, Bialystok
  - Medical Univeristy of Bialystok, Bialystok
  - Department of Cardiology and Internal Medicine, Medical University of Gdansk, Gdynia, Poland, Gdansk
- Department of Internal diseases, I.M.Sechenov First Moscow State Medical University, Moscow, Russian Federation, Moscow, Russia
- iverpool Centre for Cardiovascular Science, University of Liverpool and Liverpool Heart & Chest Hospital, Liverpool, United Kingdom, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only all IPD that underlie results in a futher publication

REFERENCES:
- [Result] Tomaszuk-Kazberuk A, Kozinski M, Kuzma L, Bujno E, Lopatowska P, Rogalska E, Dobrzycki S, Sobkowicz B, Lip GYH. Atrial fibrillation is more frequently associated with nonobstructive coronary lesions: the Bialystok Coronary Project. Pol Arch Intern Med. 2020 Dec 22;130(12):1029-1036. doi: 10.20452/pamw.15635. Epub 2020 Oct 5. PMID 33016687
- [Result] Rogalska E, Kuzma L, Wojszel ZB, Kurasz A, Napalkov D, Sokolova A, Tomaszuk-Kazberuk A. Atrial fibrillation is a predictor of nonobstructive coronary artery disease in elective angiography in old age: a cross-sectional study in Poland and Russia. Aging Clin Exp Res. 2022 Jan;34(1):175-183. doi: 10.1007/s40520-021-01895-y. Epub 2021 Jun 11. PMID 34117626